CLINICAL TRIAL: NCT02325323
Title: Prospective Cohort Study: Prognosis and Risk Factors of Gastric Cancer in Patients With Intestinal Metaplasia
Brief Title: Prognosis and Risk Factors of Gastric Cancer in Patients With Intestinal Metaplasia
Acronym: GASTRIMED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société nationale française de gastro-entérologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-DLE-GASTRIMED
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-11

CONDITIONS: Stomach Cancer
Keywords: stomach cancer; gastric intestinal metaplasia; prospective cohort; low grade dysplasia; high grade dysplasia; prognosis factor; gastric cancer risks
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy slides.
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective cohort study aims to assess the incidence of gastric cancer in patients with intestinal metaplasia in body of stomach or angular incisure.

As secondary objectives, among the patients included in the cohort, the study will:

* assess the incidence of low grade dysplasia,
* assess the incidence of high grade dysplasia in patients with low grade dysplasia,
* identify risk factors of progression to dysplasia and gastric cancer.

DETAILED DESCRIPTION:
This is a French nationwide prospective study. 2000 patients will be enrolled by 3500 gastroenterologists, either in private or public healthcare settings.

All patients will undergo an endoscopy with gastric sampling in order to biopsy:

* 1 sample each in anterior and posterior surfaces of antrum
* 1 sample in lesser curvature
* 1 sample each in anterior and posterior surfaces of body of stomach

Patients will be contacted every 12 months and followed up for 3 years by their gastroenterologist. The follow-up will be performed according to the 2012 European Guideline on Management of Precancerous Conditions and Lesions in the stomach (Endoscopy 2012, Jan; 44(1): 74-94). Patients will also receive a 6-monthly phone call from their gastroenterologist in order to know if any gastric symptom has appeared. At any time, patients should contact their gastroenterologist to inform them about new gastric symptoms.

During follow-up, the frequency of gastroscopy with biopsy depends on the stage of lesions:

* patients with intestinal metaplasia: gastroscopy at 36 months.
* patients with dysplasia: an annual gastroscopy will be performed.

In case of low grade dysplasia confirmed by pathologist at inclusion, patients will undergo 1 year later another endoscopy with gastric sampling in order to biopsy:

* 4 circumferential samplings of antrum
* 1 sampling of curvature
* 4 circumferential samplings of body of stomach

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Gastroscopic examination with biopsy in the 6 months preceding inclusion, with intestinal metaplasia in body of stomach or angular incisure.
* Patient does not oppose to participate to the study.

Exclusion Criteria:

* Progressive concomitant disease with life expectancy less than 3 years.
* Gastric cancer at the time of inclusion.
* Patient with previous oesophageal cancer.
* Patient with previous gastric surgery.
* Anticipated obstacles to follow-up during the study (e.g., understanding difficulties, homelessness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric metaplasia consulting a gastroenterologist in any private or public setting in France.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of gastric cancer or high grade dysplasia of the gastric mucosa | 3 years
  Incidence of gastric cancer or high grade dysplasia of the gastric mucosa during the 3-year follow-up.

SECONDARY OUTCOMES:
Percentage of development of low grade dysplasia | 3 years
  Percentage of development of low grade dysplasia in patients initially with intestinal metaplasia without dysplasia.
Percentage of development of gastric cancer or high grade dysplasia | 3 years
  Percentage of development in 3 years of gastric cancer or high grade dysplasia lesion, in patients initially with low grade dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LAMARQUE, MD, PhD, Principal Investigator — Hôpital Ambroise Paré, APHP
Locations (1):
- Service Hépato-gastro-Entérologie, Hôpital Ambroise Paré, Boulogne-Billancourt, Île-de-France Region, France